CLINICAL TRIAL: NCT00201968
Title: Functional Electrical Stimulation-Assisted Walking: Reduction of Secondary Complications Due to Spinal Cord Injury
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ontario Neurotrauma Foundation (Other)
Responsible Party: Principal Investigator, Milos Popovic, Senior Scientist, Toronto Rehabilitation Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REL-2004-3
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-02

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Electric Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FES training (Other): Arm 1 receives functional electrical stimulation while walking on body weight suspension training.
  Interventions: Device: Compex Motion Stimulator
- Control Group training (Other): Aerobic and resistance training program
  Interventions: Other: Conventional Exercise

INTERVENTIONS:
Device: Compex Motion Stimulator — Functional Electrical Stimulation applied to the lower limbs of SCI individuals in order to stimulate walking while on Body Weight Support Treadmill
  Other Names: Brand Name: Loko 70; Code Names: BWST, FES
  Arms: FES training
Device: Compex Motion Stimulator — Specific functional electrical stimulation program developed for each individual applied while walking on the treadmill.
  Other Names: FES, Electrical stimulation
  Arms: FES training
Other: Conventional Exercise — An aerobic and resistance training program.
  Other Names: Conventional Physiotherapy
  Arms: Control Group training

SUMMARY:
The purpose of this study is to evaluate whether an aerobic and resistance training program or a functional electrical stimulation-assisted Walking program is more effective for reducing health complications related to spinal cord injury, for example, the occurrence of bladder infections, pressure sores and/or frequency of spasms. It is hypothesized that the functional electrical stimulation-assisted walking will have a greater impact on secondary complications than the aerobic and resistance training program.

DETAILED DESCRIPTION:
A barrier to maintaining health status and active social participation in the community for individuals with spinal cord injury (SCI) is the broad number of secondary medical complications typically associated with their injury, such as bone loss, spasticity, urinary tract infections and pressure sores. Functional electrical stimulation (FES) is an intervention that applies short current pulses to muscles and causes them to contract. FES can be applied to individuals with SCI to help them restore functions such as walking and grasping by contracting groups of paralyzed muscles in an orchestrated manner. Pilot work conducted by our research group suggests that applying FES to augment functional improvement often reduces incidents of secondary complications such as spasticity, pressure sores, and swelling of the legs. Specifically, functional and meaningful walking tasks performed on a regular basis with the help of FES therapy have the potential to improve overall physical and psychological well being of persons with incomplete SCI. This study seeks to demonstrate that thrice-weekly FES training for 4 months can restore/improve walking function in chronic, incomplete SCI individuals and that this therapy will considerably reduce the occurrences of secondary complications due to SCI. This will subsequently promote opportunities for active social participation and enhance the quality of life for SCI consumers. Comparison: 32 individuals with chronic, incomplete SCI will be randomized to either thrice-weekly FES therapy OR thrice-weekly aerobic and resistance training. The study will determine which therapy is superior for improving walking function and reducing secondary complications associated with SCI after 4 months of training, and after 2-month and 8-month follow-up periods.

ELIGIBILITY:
Inclusion Criteria:

* incomplete spinal cord lesion of sudden onset between C6 and T12 that is motor incomplete (grade C or D on the ASIA neurological impairment scale). The injury must have occurred at least two years prior to recruitment

Exclusion Criteria:

* contraindications for FES, such as cardiac pacemakers, skin lesions or rush at potential electrode sites, or denervation of targeted muscles.
* pressure ulcers anywhere on the lower extremities
* hypertension that is uncontrolled
* symptoms of orthostatic hypotension when standing for 15 minutes
* susceptibility to autonomic dysreflexia, requiring medication.
* if there is a history of cardiovascular disease, participants must obtain medical clearance from their physician before inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2005-04; Primary Completion 2013-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Whole body muscle mass via dual-energy x-ray absorptiometry | Baseline, 4 month and 12 months
Bone density at different hip, spine, proximal and distal femur and proximal Tibia using dual-energy xray absorptiometry | Baseline, 4 month and 12 months
Bone density, bone geometry and muscle area via computed tomography, | Baseline, 4 month and 12 months
Spasticity via Ashworth Scale and Pendulum Test, and | Baseline, 4 months, 6 months and 12 months
Factor analysis of electromyography and kinematics of gait. | Baseline, 4months and 6 months

SECONDARY OUTCOMES:
Incidence of urinary tract infections, | Over 12 months
Spinal cord independence measure, | Baseline and 12 months
Urinary N-telopeptide and serum osteocalcin, | Baseline, 4 month, 6 month and 12 months
Timed up and go and two-minute walk test (functional mobility), | Baseline, 4 months, 6 months and 12 months
Incidence of pressure sores, | Over 12 months
Reintegration to normal living index, | Baseline, 4, 6 and 12 months
Satisfaction with life scale, | Baseline, 4 , 6 and 12 months
Instrumental Activities of Daily Living SubScale, | Baseline, 4, 6 and 12 months
Craig Handicap assessment and reporting technique, and | Baseline, 4, 6 and 12 months
client perception of treatment (qualitative). | At 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Milos Popovic, PhD, Principal Investigator — University of Toronto
Locations (1):
- Lyndhurst Centre, Toronto Rehabilitation Institute, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Kapadia N, Masani K, Catharine Craven B, Giangregorio LM, Hitzig SL, Richards K, Popovic MR. A randomized trial of functional electrical stimulation for walking in incomplete spinal cord injury: Effects on walking competency. J Spinal Cord Med. 2014 Sep;37(5):511-24. doi: 10.1179/2045772314Y.0000000263. PMID 25229735
- [Derived] Giangregorio L, Craven C, Richards K, Kapadia N, Hitzig SL, Masani K, Popovic MR. A randomized trial of functional electrical stimulation for walking in incomplete spinal cord injury: effects on body composition. J Spinal Cord Med. 2012 Sep;35(5):351-60. doi: 10.1179/2045772312Y.0000000041. PMID 23031172